CLINICAL TRIAL: NCT05071443
Title: VACuum-Assisted Closure for Necrotizing Soft Tissue infecTIONs
Acronym: VACATION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP200021
Record Dates: First submitted 2021-07-19; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-07

CONDITIONS: Necrotising Soft Tissue Infections
Keywords: Necrotising soft tissue infections; Necrotising fasciitis; Negative pressure wound therapy
MeSH Terms: conditions — Fasciitis, Necrotizing | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This committee comprises experts (a dermatologist, a plastic surgeon, and a nurse specialized in wound care) tasked with validating in a consistent manner, blinded to the randomization arm, the aspect of the primary endpoint relating to cutaneous healing, based on standard photographs taken on a weekly basis by the clinical research nurse. Photographs will be made available to members of the adjudication committee through an online platform (Dispose AP-HP) or a digital support.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative pressure wound therapy (NPWT) (Experimental): Negative pressure wound therapy (NPWT): an NPWT device will be applied hermetically from randomization to skin grafting.
  Interventions: Other: Negative pressure wound therapy (NPWT)
- Conventional dressing (Active Comparator): Conventional dressing will be performed from randomization to skin grafting. The dressings will be performed following usual procedures of investigating centers
  Interventions: Other: Conventional dressing

INTERVENTIONS:
Other: Negative pressure wound therapy (NPWT) — The therapeutic intervention being tested is the use of a negative pressure wound therapy (NPWT) device. Several medical devices are currently being used and are based on the same principle. They involve applying negative pressure, generally between -100 and -150 mmHg, to a wound using a dressing (mostly a polyurethane foam dressing with hydrophobic pores), which hermetically covers the wound's surface and is connected to a container for collecting the fluids drained off. These devices are widely available and used to treat post-operative wounds.
  Duration of treatment: the use of NPWT will be maintained until the recovery of the skin has been achieved by the skin graft. An average duration of 3 weeks' treatment is expected in the intervention group.
  Arms: Negative pressure wound therapy (NPWT)
Other: Conventional dressing — Conventional dressings will be performed from randomization to skin grafting and applied every day based on the methods normally used in the participating centres, and also until the recovery of the skin has been achieved by the skin graft.
  This generally involves local care provided on a daily basis, ensuring gentle mechanical and chemical debridement by covering the wound with alginate type or other dressings, according to the condition of the wound. The methods used to apply these conventional dressings will be recorded.
  Arms: Conventional dressing

SUMMARY:
Intro: Necrotizing and soft tissue infections (NSTI) are life-threatening bacterial infections characterized by subcutaneous tissue, fascia or muscle necrosis. The hospital mortality of NSTI is high, comprised between 20 and 30%. NSTIs represent the 4th cause of septic shock. Early management of NSTIs requires a coordinated and multidisciplinary approach, including broad-spectrum antibiotic administration, management of organ failures and aggressive surgical debridement with excision of all necrotic and infected tissues. NSTIs involve the lower limbs in about 70% of cases and lead in 15% of cases to limb amputation. During the early post-operative phase, daily wound care is required using conventional dressings. As soon as the infectious process is controlled, typically within 7 to 10 days of the initial debridement, the main goal of wound dressing is to allow for a granulation tissue to develop so that to perform a skin grafting. Negative pressure wound therapy (NPWT), which consists in applying a negative pressure on the wound surface, may be used to this effect. A dedicated dressing is connected to a device that generates a negative pressure and collects exudates. NPWT may have a positive effect on wound healing by removing exudate, increasing regional perfusion and patient comfort and reducing infections. Beneficial effects of NPWT have been suggested by case series. However, no randomized controlled trial are currently available to adequately assess its efficiency and the 2014 guidelines of the Infectious Diseases Society of America (IDSA) on NSTI did not provide recommendations regarding NPWT use for managing NSTI wounds. The study's hypothesis is that in patients managed for NSTIs, NPWT: 1) may accelerate skin grafting and complete wound healing; and 2) improve functional outcomes.

DETAILED DESCRIPTION:
Hypothesis/Objective: To demonstrate in patients who underwent a surgical debridement of the lower limb for NSTI a superiority of a wound dressing strategy using NPWT (intervention) as compared with conventional wound dressing on local healing (complete) and the recovery of walking.

Method: Open-label randomized controlled trial with blinded assessment of the primary end point. Randomization in two arms: experimental group (NPWT) versus control group (conventional dressing) until skin grafting (decided by the attending surgeon).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written informed consent
* NSTI/NF of the lower limb clinically suspected and confirmed by surgery with a first debridement performed since 5 days or more
* Infection considered controlled (i.e., no more surgical debridement is necessary)
* Last debridement performed at least 72 hours before
* Affiliation to a social security system

Exclusion Criteria:

* Limited life expectancy
* NPWT already initiated for the current NSTI/NF episode
* 1st surgical debridement performed less than 5 days or more than 15 days before
* High risk of bleeding (blood vessels exposed)
* Local neoplasia
* Risk of organ or peripheral nerve injury
* Impossibility to set up a NPWT dressing hermetically
* Limb amputation
* Patient unable to walk without help
* Women who are pregnant or are breast-feeding, or are of childbearing age and do not use or do not plan to use acceptable birth control measures
* Patients under legal protection
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The time elapsed between randomization and the onset of a combined outcome measure including a complete healing of the diseased limb and the recovery of walking. | between Day 0 and 3 months
  Complete healing of the diseased limb is defined by more than 90% of functional skin covering the wound and Recovery of walking is defined by the ability to walk at least 100 steps, corresponding to approximately 30 meters, without help

SECONDARY OUTCOMES:
Activities of Daily Living score | at Day 0, 3 months and 6 months
Short Form - 36 | at Day 0, 3 months and 6 months
Pain assessment | between Day 0 and 3 months
  Pain assessment at each wound care by the patient (visual analogic scale), the nurse (behavioral pain scale) and quantification of morphine consumption (in morphine base equivalent): measured by the investigator at each wound care
Quantification of the number of anesthesia procedures (general anesthesia, sedation) | between Day 0 and 6 months
Time elapsed between randomization and skin grafting | between Day 0 and 6 months
Number of local superinfection episodes | between Day 0 and 3 months
Quantification of the walking capacity | at 3 months and 6 months
  measured over one week with a pedometer by the research nurse, at 3 and 6 months
Duration of hospital stay | between Day 0 and 6 months
Quantification of the time needed for each wound care before randomization and skin grafting | between Day 0 and 6 months
  this measure will be recorded once a week for one wound care
Need for stopping the NPWT | between Day 0 and 3 months
Number of surgeries performed between randomization and skin grafting | between Day 0 and 6 months
  All surgeries will be recorded, including their date and indication
Number of surgeries performed after skin grafting | between Day 0 and 6 months
  All surgeries will be recorded, including their date and indication, all surgeries will be recorded, including their date and indication
Mortality assessed | at 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas DE PROST, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU Henri Mondor, Créteil, France